CLINICAL TRIAL: NCT04116944
Title: Effects of Resistance Exercise Among Young Adults With and Without Analogue Generalized Anxiety Disorder: A Protocol for a Randomized Controlled Trial
Brief Title: The Resistance Exercise Training for Worry Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Collaborators: Irish Research Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017_03_18_EHS
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Analogue Generalized Anxiety Disorder
Keywords: anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Resistance Training; Waiting Lists

STUDY DESIGN:
Intervention Model Description: Two parallel, randomized controlled trials of an eight-week resistance exercise training intervention compared to a wait-list control condition among young adults with and without analogue-Generalized Anxiety Disorder
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principal investigator was blinded to participant allocation, and the analyses were performed blinded to group. Participants' individual identification numbers assigned at baseline were used during the course of the trial. Following full data extraction from SurveyMonkey.com, identifying information were removed, such that no participant could be identified in the working dataset through one, or a combination of different variables.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Analogue-Generalized Anxiety Disorder Resistance Training (Experimental): Resistance exercise training among young adults with analogue-Generalized Anxiety Disorder
  Interventions: Behavioral: Resistance exercise training
- Analogue-Generalized Anxiety Disorder Wait-List (Other): 8-week wait-list control condition among young adults with analogue-Generalized Anxiety Disorder
  Interventions: Other: Wait-list
- Non-Analogue-Generalized Anxiety Disorder Resistance Training (Experimental): Resistance exercise training among young adults without analogue-Generalized Anxiety Disorder
  Interventions: Behavioral: Resistance exercise training
- Non-Analogue-Generalized Anxiety Disorder Wait-List (Other): 8-week wait-list control condition among young adults with analogue-Generalized Anxiety Disorder
  Interventions: Other: Wait-list

INTERVENTIONS:
Behavioral: Resistance exercise training — The ecologically-valid resistance exercise training was designed according to World Health Organization and American College of Sports Medicine guidelines. The eight-week, twice-weekly intervention was designed to be performed at a moderate intensity. The resistance of each exercise was such that when participants could successfully complete 2 sets of 12 repetitions at a certain load, the resistance was increased incrementally up to 5% for the following session. Exercise sessions were scheduled with at least one day of rest between sessions. The eight exercises included the barbell squat, barbell bench press, hexagon bar deadlift, dumbbell shoulder lateral raise, barbell bent over rows, dumbbell lunges, dumbbell curls, and abdominal crunches.
  Other Names: weight-lifting; strength training
  Arms: Analogue-Generalized Anxiety Disorder Resistance Training; Non-Analogue-Generalized Anxiety Disorder Resistance Training
Other: Wait-list — Participants randomized to the delayed-start wait-list condition completed questionnaires once-weekly. The investigator sent a weekly email to the participant providing links to the questionnaires. Participants that completed the eight-week wait-list condition were offered the eight weeks of RET either immediately upon completion, or later at a time of their convenience while the trial was ongoing. Each participant randomized to the eight-week wait-list also completed two 30-minute bouts of seated quiet rest in an empty room at weeks one and eight.
  Arms: Analogue-Generalized Anxiety Disorder Wait-List; Non-Analogue-Generalized Anxiety Disorder Wait-List

SUMMARY:
This protocol details the full methods of two parallel, randomized controlled trials of an eight-week resistance exercise training intervention compared to a wait-list control condition among young adults with and without analogue-Generalized Anxiety Disorder.

DETAILED DESCRIPTION:
Recent meta-analyses support the chronic anxiolytic effects of resistance exercise training among women with diagnosed Generalized Anxiety Disorder. However, the effects of resistance exercise training among those with subclinical, or analogue-Generalized Anxiety Disorder is unknown. This protocol details the full methods of two parallel, randomized controlled trials of an eight-week resistance exercise training intervention compared to a wait-list control condition among young adults with and without analogue-Generalized Anxiety Disorder. Analogue-Generalized Anxiety Disorder status was determined using validated cut-scores for both the Psychiatric Diagnostic Screening Questionnaire Generalized Anxiety Disorder sub-scale score of 6 or greater, and the Penn State Worry Questionnaire score of 45 or greater. The ecologically-valid resistance exercise training was designed according to World Health Organization and American College of Sports Medicine guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were age 18-40y; no medical contraindication to safe participation in resistance exercise training; and no current pregnancy or lactation.

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
Analogue-Generalized Anxiety Disorder Status | Baseline
  The Psychiatric Diagnostic Screening Questionnaire Generalized Anxiety Disorder subscale score of 6 or greater (Zimmerman & Mattia, 2001, Arch of Gen Psychiatr)
Analogue-Generalized Anxiety Disorder Status | week1
  The Psychiatric Diagnostic Screening Questionnaire Generalized Anxiety Disorder subscale score of 6 or greater (Zimmerman & Mattia, 2001, Arch of Gen Psychiatr)
Analogue-Generalized Anxiety Disorder Status | week 4
  The Psychiatric Diagnostic Screening Questionnaire Generalized Anxiety Disorder subscale score of 6 or greater (Zimmerman & Mattia, 2001, Arch of Gen Psychiatr)
Analogue-Generalized Anxiety Disorder Status | week 8
  The Psychiatric Diagnostic Screening Questionnaire Generalized Anxiety Disorder subscale score of 6 or greater (Zimmerman & Mattia, 2001, Arch of Gen Psychiatr)
Analogue-Generalized Anxiety Disorder Status | Baseline
  The Penn State Worry Questionnaire score of 45 or greater (Meyer et al., 1990, Behav Res and Ther)
Analogue-Generalized Anxiety Disorder Status | week1
  The Penn State Worry Questionnaire score of 45 or greater (Meyer et al., 1990, Behav Res and Ther)
Analogue-Generalized Anxiety Disorder Status | week 4
  The Penn State Worry Questionnaire score of 45 or greater (Meyer et al., 1990, Behav Res and Ther)
Analogue-Generalized Anxiety Disorder Status | week 8
  The Penn State Worry Questionnaire score of 45 or greater (Meyer et al., 1990, Behav Res and Ther)

SECONDARY OUTCOMES:
Anxiety Symptoms | Baseline
  State and trait anxiety were measured using the State (STAI-Y1) and Trait (STAI-Y2) subscales of the State-Trait Anxiety Inventory (Spielberger, 2010, Corsini Encycl of Psychol)
Anxiety Symptoms | week 1
  State and trait anxiety were measured using the State (STAI-Y1) and Trait (STAI-Y2) subscales of the State-Trait Anxiety Inventory (Spielberger, 2010, Corsini Encycl of Psychol)
Anxiety Symptoms | week 2
  State and trait anxiety were measured using the State (STAI-Y1) and Trait (STAI-Y2) subscales of the State-Trait Anxiety Inventory (Spielberger, 2010, Corsini Encycl of Psychol)
Anxiety Symptoms | week 3
  State and trait anxiety were measured using the State (STAI-Y1) and Trait (STAI-Y2) subscales of the State-Trait Anxiety Inventory (Spielberger, 2010, Corsini Encycl of Psychol)
Anxiety Symptoms | week 4
  State and trait anxiety were measured using the State (STAI-Y1) and Trait (STAI-Y2) subscales of the State-Trait Anxiety Inventory (Spielberger, 2010, Corsini Encycl of Psychol)
Anxiety Symptoms | week 5
  State and trait anxiety were measured using the State (STAI-Y1) and Trait (STAI-Y2) subscales of the State-Trait Anxiety Inventory (Spielberger, 2010, Corsini Encycl of Psychol)
Anxiety Symptoms | Week 6
  State and trait anxiety were measured using the State (STAI-Y1) and Trait (STAI-Y2) subscales of the State-Trait Anxiety Inventory (Spielberger, 2010, Corsini Encycl of Psychol)
Anxiety Symptoms | Week 7
  State and trait anxiety were measured using the State (STAI-Y1) and Trait (STAI-Y2) subscales of the State-Trait Anxiety Inventory (Spielberger, 2010, Corsini Encycl of Psychol)
Anxiety Symptoms | Week 8
  State and trait anxiety were measured using the State (STAI-Y1) and Trait (STAI-Y2) subscales of the State-Trait Anxiety Inventory (Spielberger, 2010, Corsini Encycl of Psychol)
Depressive Symptoms | Baseline
  16-item Quick Inventory of Depressive Symptomatology (Rush et al., 2003, Bio Psychiatr)
Depressive Symptoms | Week 1
  16-item Quick Inventory of Depressive Symptomatology (Rush et al., 2003, Bio Psychiatr)
Depressive Symptoms | Week 2
  16-item Quick Inventory of Depressive Symptomatology (Rush et al., 2003, Bio Psychiatr)
Depressive Symptoms | Week 3
  16-item Quick Inventory of Depressive Symptomatology (Rush et al., 2003, Bio Psychiatr)
Depressive Symptoms | Week 4
  16-item Quick Inventory of Depressive Symptomatology (Rush et al., 2003, Bio Psychiatr)
Depressive Symptoms | Week 5
  16-item Quick Inventory of Depressive Symptomatology (Rush et al., 2003, Bio Psychiatr)
Depressive Symptoms | Week 6
  16-item Quick Inventory of Depressive Symptomatology (Rush et al., 2003, Bio Psychiatr)
Depressive Symptoms | Week 7
  16-item Quick Inventory of Depressive Symptomatology (Rush et al., 2003, Bio Psychiatr)
Depressive Symptoms | Week 8
  16-item Quick Inventory of Depressive Symptomatology (Rush et al., 2003, Bio Psychiatr)
Mood | Baseline
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Mood | Week 1
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Mood | Week 2
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Mood | Week 3
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Mood | Week 4
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Mood | Week 5
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Mood | Week 6
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Mood | Week 7
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Mood | Week 8
  Subscales of the Profile of Mood States - Brief Form (McNair et al., 1992)
Irritability | Baseline
  21-item Irritability Questionnaire (Craig et al., 2008, Psychiatr Res)
Irritability | Week 1
  21-item Irritability Questionnaire (Craig et al., 2008, Psychiatr Res)
Irritability | Week 2
  21-item Irritability Questionnaire (Craig et al., 2008, Psychiatr Res)
Irritability | Week 3
  21-item Irritability Questionnaire (Craig et al., 2008, Psychiatr Res)
Irritability | Week 4
  21-item Irritability Questionnaire (Craig et al., 2008, Psychiatr Res)
Irritability | Week 5
  21-item Irritability Questionnaire (Craig et al., 2008, Psychiatr Res)
Irritability | Week 6
  21-item Irritability Questionnaire (Craig et al., 2008, Psychiatr Res)
Irritability | Week 7
  21-item Irritability Questionnaire (Craig et al., 2008, Psychiatr Res)
Irritability | Week 8
  21-item Irritability Questionnaire (Craig et al., 2008, Psychiatr Res)
Sleep Quality | Baseline
  Pittsburgh Sleep Quality Index (Buysse et al., 1989, Psychiatr Res)
Sleep Quality | Week 1
  Pittsburgh Sleep Quality Index (Buysse et al., 1989, Psychiatr Res)
Sleep Quality | Week 2
  Pittsburgh Sleep Quality Index (Buysse et al., 1989, Psychiatr Res)
Sleep Quality | Week 3
  Pittsburgh Sleep Quality Index (Buysse et al., 1989, Psychiatr Res)
Sleep Quality | Week 4
  Pittsburgh Sleep Quality Index (Buysse et al., 1989, Psychiatr Res)
Sleep Quality | Week 5
  Pittsburgh Sleep Quality Index (Buysse et al., 1989, Psychiatr Res)
Sleep Quality | Week 6
  Pittsburgh Sleep Quality Index (Buysse et al., 1989, Psychiatr Res)
Sleep Quality | Week 7
  Pittsburgh Sleep Quality Index (Buysse et al., 1989, Psychiatr Res)
Sleep Quality | Week 8
  Pittsburgh Sleep Quality Index (Buysse et al., 1989, Psychiatr Res)
Non-Intervention Physical Activity | Baseline
  7-day Physical Activity Recall (Blair et al., 1985, Am J of Epidemiol)
Non-Intervention Physical Activity | Week 1
  7-day Physical Activity Recall (Blair et al., 1985, Am J of Epidemiol)
Non-Intervention Physical Activity | Week 2
  7-day Physical Activity Recall (Blair et al., 1985, Am J of Epidemiol)
Non-Intervention Physical Activity | Week 3
  7-day Physical Activity Recall (Blair et al., 1985, Am J of Epidemiol)
Non-Intervention Physical Activity | Week 4
  7-day Physical Activity Recall (Blair et al., 1985, Am J of Epidemiol)
Non-Intervention Physical Activity | Week 5
  7-day Physical Activity Recall (Blair et al., 1985, Am J of Epidemiol)
Non-Intervention Physical Activity | Week 6
  7-day Physical Activity Recall (Blair et al., 1985, Am J of Epidemiol)
Non-Intervention Physical Activity | Week 7
  7-day Physical Activity Recall (Blair et al., 1985, Am J of Epidemiol)
Non-Intervention Physical Activity | Week 8
  7-day Physical Activity Recall (Blair et al., 1985, Am J of Epidemiol)
A novel questionnaire assessing expectancy of exercise to improve or not to improve physical and mental health outcomes. (Lindheimer et al., 2019, Eur J of Sport Sci) | Baseline
  Participants are asked to what degree they believe a single bout of exercise will improve or worsen various domains of physical and mental health
A novel questionnaire assessing expectancy of exercise to improve or not to improve physical and mental health outcomes. (Lindheimer et al., 2019, Eur J of Sport Sci) | Week 1
  Participants are asked to what degree they believe a single bout of exercise will improve or worsen various domains of physical and mental health
A novel questionnaire assessing expectancy of exercise to improve or not to improve physical and mental health outcomes. (Lindheimer et al., 2019, Eur J of Sport Sci) | Week 2
  Participants are asked to what degree they believe a single bout of exercise will improve or worsen various domains of physical and mental health
A novel questionnaire assessing expectancy of exercise to improve or not to improve physical and mental health outcomes. (Lindheimer et al., 2019, Eur J of Sport Sci) | Week 3
  Participants are asked to what degree they believe a single bout of exercise will improve or worsen various domains of physical and mental health
A novel questionnaire assessing expectancy of exercise to improve or not to improve physical and mental health outcomes. (Lindheimer et al., 2019, Eur J of Sport Sci) | Week 4
  Participants are asked to what degree they believe a single bout of exercise will improve or worsen various domains of physical and mental health
A novel questionnaire assessing expectancy of exercise to improve or not to improve physical and mental health outcomes. (Lindheimer et al., 2019, Eur J of Sport Sci) | Week 5
  Participants are asked to what degree they believe a single bout of exercise will improve or worsen various domains of physical and mental health
A novel questionnaire assessing expectancy of exercise to improve or not to improve physical and mental health outcomes. (Lindheimer et al., 2019, Eur J of Sport Sci) | Week 6
  Participants are asked to what degree they believe a single bout of exercise will improve or worsen various domains of physical and mental health
A novel questionnaire assessing expectancy of exercise to improve or not to improve physical and mental health outcomes. (Lindheimer et al., 2019, Eur J of Sport Sci) | Week 7
  Participants are asked to what degree they believe a single bout of exercise will improve or worsen various domains of physical and mental health
A novel questionnaire assessing expectancy of exercise to improve or not to improve physical and mental health outcomes. (Lindheimer et al., 2019, Eur J of Sport Sci) | Week 8
  Participants are asked to what degree they believe a single bout of exercise will improve or worsen various domains of physical and mental health
Attentional Biases | Baseline
  Attentional bias to positive, negative, and neutral facial images (Gotlin et al., 2004, J of Abnorm Psychol)
Attentional Biases | Week 1
  Attentional bias to positive, negative, and neutral facial images (Gotlin et al., 2004, J of Abnorm Psychol)
Attentional Biases | Week 8
  Attentional bias to positive, negative, and neutral facial images (Gotlin et al., 2004, J of Abnorm Psychol)
Cognitive Function | Baseline
  Stroop colour and word test, (Williams et al., 1996, Psychol Bull) and Trail Making Test (Tombaugh, 2004, Arch of Clin Neuropsychol)
Cognitive Function | Week1
  Stroop colour and word test, (Williams et al., 1996, Psychol Bull) and Trail Making Test (Tombaugh, 2004, Arch of Clin Neuropsychol)
Cognitive Function | Week 8
  Stroop colour and word test, (Williams et al., 1996, Psychol Bull) and Trail Making Test (Tombaugh, 2004, Arch of Clin Neuropsychol)

CONTACTS AND LOCATIONS:
Locations (1):
- The Department of Physical Education and Sport Sciences Building, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcomes measures will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Primary outcome data will be made available for five years at six months following publication of primary outcome summary data. Secondary outcome data will be made available for five years at six months following publications of secondary outcome summary data.
Access Criteria: Proposals should be directed to matthew.herring@ul.ie. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] O'Sullivan D, Gordon BR, Lyons M, Meyer JD, Herring MP. Effects of Resistance Exercise on Depressed Mood State: A Randomized Controlled Trial. Med Sci Sports Exerc. 2025 Nov 1;57(11):2496-2502. doi: 10.1249/MSS.0000000000003769. Epub 2025 May 29. PMID 40440519
- [Derived] Gordon BR, McDowell CP, Lyons M, Herring MP. The effects of acute resistance exercise among young adults: A randomized controlled trial. J Affect Disord. 2022 Feb 15;299:102-107. doi: 10.1016/j.jad.2021.11.049. Epub 2021 Nov 18. PMID 34801607
- [Derived] Gordon BR, McDowell CP, Lyons M, Herring MP. Resistance exercise training for anxiety and worry symptoms among young adults: a randomized controlled trial. Sci Rep. 2020 Oct 16;10(1):17548. doi: 10.1038/s41598-020-74608-6. PMID 33067493